CLINICAL TRIAL: NCT00896714
Title: Impact of Environmental and Demographic Factors on Pre-operative Doses of Anesthetic Agents (Prospective Multicenter Study)
Brief Title: Factors Influencing Anesthetic Drug Requirement
Acronym: PosoAnes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008/44
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Closed loop anesthesia (Experimental)
  Interventions: Device: Closed loop anesthesia

INTERVENTIONS:
Device: Closed loop anesthesia — Propofol and Remifentanil are administered automatically using a closed-loop system

SUMMARY:
The main objective of the study is to analyze the influence of several environmental (i.e., timing: seasonal, circadian) and demographic conditions (i.e., age, gender, menstrual cycle) on anesthetic drug requirements (hypnotic and opiate).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled surgery under general anesthesia, agreeing to participate in the study

Exclusion Criteria:

* Age under 18 years
* Pregnancy, breastfeeding woman
* Allergy to propofol, soybeans or peanuts
* Allergy to sufentanil, remifentanil, morphine,
* Allergy to a muscle relaxant or to any of its excipients
* Known hypersensitivity to sufentanil, remifentanil, or to other derivates of fentanyl
* History of central neurological disorder or brain injury
* Patient with dementia
* Patient with pacemaker
* Patient receiving psychotropic drugs or morphine agonist-antagonists
* Surgery on the skull and/or operating position preventing the use of a bispectral index sensor in suitable conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3278 (Actual)
Dates: Start 2009-05-04 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
The dose of propofol required to maintain BIS (bispectral index) between 40 and 60 during maintenance of anesthesia | during anesthesia

SECONDARY OUTCOMES:
Propofol dose required for anesthesia induction | intraoperative period
Remifentanil dose required for anesthesia induction | intraoperative period
Remifentanil dose requirements for maintenance of anesthesia | intraoperative period
Wake up time | intraoperative period
Explicit memorisation | post-operative period
Propofol and remifentanil requirements according to the surgical technique | post-operative period
Analysis of subgroup of patients according to their clinical status | post-operative period
  analysis of subgroup of patients according to their clinical status (eg: age)
Analysis of subgroup of patients according to the surgical approach | post-operative period
  analysis of subgroup of patients according to the surgical approach ("open" surgery versus "minimal invasive" surgery)
Analysis of subgroup of patients according to their pathology | post-operative period
  analysis of subgroup of patients according to their pathology (eg: burns)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (4):
- France (4):
  - CHU Besançon, Besançon
  - Centre Hospitalier de Dreux, Dreux
  - Hôpital Tenon, Paris
  - Hôpital Foch, Suresnes